CLINICAL TRIAL: NCT06425146
Title: Clinical-biological, Prospective, Monocentric Cohort Study to Describe Somatic Mutations in Healthy Oral Mucosa From Patients With Oral Squamous Cell Carcinoma (OSCC)
Brief Title: Tobacco, Alcohol and Cancerization of the Oral Mucosa (TACO)
Acronym: TACO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ET23-384 TACO
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-05

CONDITIONS: Oral Squamous Cell Carcinomas
Keywords: Somatic mutations; Healthy oral mucosa; oral cancer; OSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: A clinical-biological cohort of patients with epidermoid carcinomas of the oral cavity.
  Blood sample and cytobrush sample at inclusion and before anti-cancer treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical-biological cohort (Other): A clinical-biological cohort of 30 patients with epidermoid carcinomas of the oral cavity.
  Blood sample and cytobrush sample at inclusion and before anti-cancer treatment.
  Interventions: Procedure: Cytobrush sample; Procedure: Blood sampling

INTERVENTIONS:
Procedure: Cytobrush sample — Healthy oral mucosa will be collected using a cytobrush, which is a minimally invasive method for patients
Procedure: Blood sampling — Blood sampling (6 mL), taken from a routine biological exam

SUMMARY:
The goal of this project is to describe somatic mutations of healthy oral mucosa from patients with oral squamous cell carcinoma (OSCC).

DETAILED DESCRIPTION:
Epidermoid carcinomas of upper aerodigestive tract are the 8th most common cancers in the world. Worldwide, this represents more than 500.000 cases per year and 20.000 cases per year in France (statistics 2018-2020). Among these cancers, oral squamous cell carcinoma (OSCC) are the most common location, leading to significant morbidity and mortality.

Despite recent advances in diagnosis, treatment and monitoring, the overall 5-year survival rate of patients with epidermoid carcinomas of upper aerodigestive tract has not improved significantly and remains around 40-50 % for all combined locations. These pejorative survival rates, as well as the increase in the incidence of these cancers, have not changed much over the past 30 years. This situation can be attributed in part to a diagnosis too late. Indeed, only 1/3 of patients with high-risk squamous cell carcinoma of the head and neck are diagnosed at an early stage. This issue of early diagnosis is mainly due to the lack of suitable screening and diagnostic biomarkers. Beyond diagnosis, the identification of biomarkers is also a prognostic and predictive interest since they could predict the course of the disease as well as the response to treatment.

"Drivers" mutations, with oncogenic potential, can be present from the very early stages of epidermoid carcinomas of upper aerodigestive tract and therefore constitute potential biomarkers. However, recent studies have demonstrated the presence of driver mutations in different types of oral cavity's healthy tissue, some being even associated with a protective effect against tumor initiation. In order to improve prevention and early diagnosis of OSCC, it is important to better understand the evolutionary dynamics of somatic mutations in the oral mucosa, which is still poorly characterized.

ELIGIBILITY:
Inclusion Criteria:

* I1. Male or female aged 18 years or older at the date of signature of the informed consent to participate.
* I2. Patient with histological diagnosis of epidermoid carcinomas of the oral cavity NB: All grades are eligible.
* I3. Patient naive of any systemic anti-cancer treatment (radio- or chemotherapy).
* I4. Patient able to understand, sign and date informed consent before the start of any study protocol procedure.
* I5. Patient affiliated or covered by a medical insurance

Exclusion Criteria:

* E1. Patients at high risk of bleeding, such as those on anticoagulant or antiplatelet aggregant treatment, with clotting disorders or a history of severe bleeding in the two weeks prior to inclusion.
* E2. Patient with lesions of all types on the mucosa of the cheek located on the opposite side of the area affected by an epidermoid carcinoma of the oral cavity which prevents painless removal of the healthy mucosa.
* E3. Patient who had surgery for their epidermoid carcinoma of the oral cavity more than 6 months ago.
* E4. Patient who uses cannabis.
* E5. Patient with another active tumor or HPV-positive tumors.
* E6. Patient under guardianship or curatorship or placed under the protection of justice.
* E7. Pregnant and/or nursing patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Identify somatic mutations of the driver genes from healthy oral mucosa from patients with epidermoid carcinomas of the upper aerodigestive tract | 1 year
  Identified mutations described by type and number

SECONDARY OUTCOMES:
Correlation between tobacco consumption and the total number of somatic mutations detected in the healthy oral mucosa in patients with OSCC | 1 year
  Correlation between tobacco consumption and total number of somatic mutations detected
Correlation between alcohol consumption and the total number of somatic mutations detected in the healthy oral mucosa in patients with OSCC | 1 year
  Correlation between alcohol consumption and total number of somatic mutations

OTHER OUTCOMES:
Selective advantage of OSCC driver mutations in normal-looking mucosa | 1 year
  Selective advantage of the 62 driver genes already identified
Non-drivers OSCC genes under positive selection in normal looking mucosa | 1 year
  Selective advantage of non-driver OSCC genes

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Zrounba, M.D., Principal Investigator — philippe.zrounba@lyon.unicancer.fr
Locations (1):
- Centre Léon Bérard, Lyon, France